CLINICAL TRIAL: NCT01932996
Title: Enhancing Smoking Cessation in the Homeless Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1307M39761; 2R01HL081522-05A1 (NIH)
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Cigarette Smoking; Tobacco Smoking; Smoking, Tobacco
Keywords: Smoking Cessation; Smoking Cessation Products; Tobacco Use Cessation Products
MeSH Terms: conditions — Cigarette Smoking; Tobacco Smoking; Smoking Cessation | interventions — Tobacco Use Cessation Devices; Ethanol; Methods; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated Intensive Smoking + Alcohol (Active Comparator): IS+A: 12-week treatment with nicotine patch plus nicotine gum/lozenge. An integrated intensive smoking along with an intensive alcohol intervention covering smoking cessation + alcohol abstinence using cognitive behavioral therapy, CBT, and will include weekly individual sessions for 3 months followed by study data collection visits for 3 months.
  Interventions: Drug: nicotine patch plus nicotine gum/lozenge; Behavioral: Intensive Alcohol Intervention
- Usual Care (Placebo Comparator): UC: 12-week treatment with nicotine patch plus nicotine gum/lozenge along with a one time brief smoking cessation and brief alcohol counseling both based on the USPHS's Guidelines
  Interventions: Drug: nicotine patch plus nicotine gum/lozenge

INTERVENTIONS:
Drug: nicotine patch plus nicotine gum/lozenge — 12-week treatment with nicotine patch plus nicotine gum/lozenge
  Other Names: NRT
Behavioral: Intensive Alcohol Intervention — Intensive alcohol abstinence counseling using CBT will include weekly individual sessions for 3 months followed by monthly booster group sessions for 3 months
  Other Names: Cognitive Behavioral Therapy, CBT
  Arms: Integrated Intensive Smoking + Alcohol

SUMMARY:
The goal of this research study is to enhance smoking cessation rates for homeless smokers. The original study design proposed to test the effects of 1) an Intensive Smoking Intervention, and 2) integrating alcohol abuse treatment with smoking cessation We will utilize a 3-group randomized design to test study hypotheses. The three study conditions are 1) Integrated Intensive Smoking plus Alcohol intervention using cognitive behavioral therapy (CBT), CBT-(IS+A); 2) Intensive Smoking Intervention using CBT-(IS); or 3) Usual Care (brief smoking cessation and brief alcohol counseling both based on the United States Public Health Service's Guidelines)-(UC). Due to low enrollment because of the addition of an alcohol use screening criteria, the study was changed to a two arm study and the study time frame changed. The two study conditions are 1) Integrated Intensive Smoking plus Alcohol intervention using cognitive behavioral therapy (CBT), CBT-(IS+A) and 2) Usual Care (brief smoking cessation and brief alcohol counseling both based on the United States Public Health Service's Guidelines)-(UC). The study length is reduced to 26 weeks from 52 weeks. All participants will receive 12-week treatment with nicotine patch plus nicotine gum/lozenge. Counseling will follows the protocol used in a recent study of alcohol dependent smokers and will include weekly individual sessions for 3 months followed by study data collection visits 3 months. Both study conditions will have equal number of study contacts. Study staff will make retention contacts with participants in the community during weeks that do not have study visits scheduled. Primary smoking outcome is cotinine-verified 7-day smoking abstinence at week 26 follow-up while secondary outcome is prolonged smoking abstinence at weeks 12, 16, and 26. Secondary alcohol outcome will be self-reported continuous alcohol abstinence for 90 days at week 26. Recruitment and retention will be enhanced by use of gift cards, bus passes, other non-monetary incentives, attractive intervention materials, collaboration with homeless shelters, and advice from a Community Advisory Board. Participants will be enrolled from homeless shelters and facilities in the 7-county greater Minneapolis/St. Paul metro area. Our power calculation indicates that a sample size of 215 per study condition is needed to detect proposed treatment effects.

DETAILED DESCRIPTION:
To achieve the study goal, we have selected a 3-group randomized clinical trial (RCT) design that includes 1) Usual Care, 2) Intensive smoking cessation, and 3) Integrated Intensive Smoking and Alcohol Intervention. Due to low enrollment because of the addition of an alcohol use screening criteria, the study was changed to a two arm study and the study time frame changed. The two study conditions are 1) Integrated Intensive Smoking plus Alcohol intervention using cognitive behavioral therapy (CBT), CBT-(IS+A) and 2) Usual Care (brief smoking cessation and brief alcohol counseling both based on the United States Public Health Service's Guidelines)-(UC). The study length is reduced to 26 weeks from 52 weeks. Having alcohol treatment added to the smoking intervention will enable us assess whether addressing alcohol abuse will result in improved smoking abstinence, an important scientific question that has never been studied in homeless populations.

Study conditions: Both study conditions have identical number of contacts; we considered a design in which the duration of counseling in the UC will be identical to those in the IS+A condition but decided against this because it will create a usual care condition that exceeds standard practice for brief interventions. We understand that testing hypothesis 3 confounds contact time with treatment content, and hence we will not be able to determine that observed differences in outcome are due to specific treatment components. However, given the current state of knowledge about treating homeless alcohol abusing smokers, we believe it is sufficient to show that our intervention led to improved outcome in this group without knowing if the finding is due to specific intervention content. Subsequent research will be needed to disentangle various intervention components.

All participants will receive 12-week treatment with nicotine patch plus nicotine gum/lozenge. Counseling will include weekly individual sessions for 3 months followed by study data collection visits for 3 months. Each participant will be randomly assigned to a condition, which will dictate their treatment. Each participant will be asked to engage in the therapy assigned to their condition, and work to quit smoking and consuming alcohol over a period of one year.

ELIGIBILITY:
Inclusion Criteria:

* Currently Homeless
* Smoked at least 100 cigarettes in lifetime
* AUDIT score of > or equal to 5, < or equal to 26
* Aged 18 years or older
* Willing to attend study sessions and follow other study protocol

Exclusion Criteria:

* Use of smoking cessation medications or interventions in last 30 days
* Unstable medical illness that requires immediate medical care
* AUDIT score of < 5 or > 26
* Pregnancy or other Nicotine Replacement Therapy (NRT) contraindications
* Current history or in past 6 months of psychotic disorder or major depressive disorders that is not stable on treatment for past 3 months
* Cognitive impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2015-01; Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pratt Rebekah, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Kalman D. Smoking cessation treatment for substance misusers in early recovery: a review of the literature and recommendations for practice. Subst Use Misuse. 1998 Aug;33(10):2021-47. doi: 10.3109/10826089809069815. PMID 9744841
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Rost K, Burnam MA, Smith GR. Development of screeners for depressive disorders and substance disorder history. Med Care. 1993 Mar;31(3):189-200. doi: 10.1097/00005650-199303000-00001. PMID 8450677
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- [Background] Katzman R, Brown T, Fuld P, Peck A, Schechter R, Schimmel H. Validation of a short Orientation-Memory-Concentration Test of cognitive impairment. Am J Psychiatry. 1983 Jun;140(6):734-9. doi: 10.1176/ajp.140.6.734. PMID 6846631
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Etter JF, Bergman MM, Humair JP, Perneger TV. Development and validation of a scale measuring self-efficacy of current and former smokers. Addiction. 2000 Jun;95(6):901-13. doi: 10.1046/j.1360-0443.2000.9569017.x. PMID 10946439
- [Background] DiClemente CC, Carbonari JP, Montgomery RP, Hughes SO. The Alcohol Abstinence Self-Efficacy scale. J Stud Alcohol. 1994 Mar;55(2):141-8. doi: 10.15288/jsa.1994.55.141. PMID 8189734
- [Background] Roski J, Schmid LA, Lando HA. Long-term associations of helpful and harmful spousal behaviors with smoking cessation. Addict Behav. 1996 Mar-Apr;21(2):173-85. doi: 10.1016/0306-4603(95)00047-x. PMID 8730519
- [Background] Amodei N, Lamb RJ. Convergent and concurrent validity of the Contemplation Ladder and URICA scales. Drug Alcohol Depend. 2004 Mar 8;73(3):301-6. doi: 10.1016/j.drugalcdep.2003.11.005. PMID 15036552
- [Background] Biener L, Abrams DB. The Contemplation Ladder: validation of a measure of readiness to consider smoking cessation. Health Psychol. 1991;10(5):360-5. doi: 10.1037//0278-6133.10.5.360. PMID 1935872
- [Background] Cornoni-Huntley J, Brock D, Ostfeld A, Taylor J, Wallace R. Established populations for for epidemiologic studies of the elderly: Resource data book. Washington, DCL US Department of Health and Human Services; 1986.
- [Background] Barnes LL, Mendes de Leon CF, Bienias JL, Evans DA. A longitudinal study of black-white differences in social resources. J Gerontol B Psychol Sci Soc Sci. 2004 May;59(3):S146-53. doi: 10.1093/geronb/59.3.s146. PMID 15118020
- [Background] Cohen S, Mermelstein R, Kamarck T, Hoberman H, eds. Mesuring the functional components of social support. In Sarason IG, Sarason BR, eds. Social Support: Theory, Research, and Application. The Hague, the Netherlands: Martunus Nijhoff; 1985.
- [Background] Cohen S, Lichtenstein E. Partner behaviors that support quitting smoking. J Consult Clin Psychol. 1990 Jun;58(3):304-9. doi: 10.1037//0022-006x.58.3.304. PMID 2365893
- [Background] Murray RP, Connett JE, Lauger GG, Voelker HT. Error in smoking measures: effects of intervention on relations of cotinine and carbon monoxide to self-reported smoking. The Lung Health Study Research Group. Am J Public Health. 1993 Sep;83(9):1251-7. doi: 10.2105/ajph.83.9.1251. PMID 8363000
- [Background] Cummings SR, Richard RJ. Optimum cutoff points for biochemical validation of smoking status. Am J Public Health. 1988 May;78(5):574-5. doi: 10.2105/ajph.78.5.574. PMID 3354745
- [Background] McDonell MG, Howell DN, McPherson S, Cameron JM, Srebnik D, Roll JM, Ries RK. Voucher-based reinforcement for alcohol abstinence using the ethyl-glucuronide alcohol biomarker. J Appl Behav Anal. 2012 Spring;45(1):161-5. doi: 10.1901/jaba.2012.45-161. PMID 22403460
- [Background] Bernard R. Research Methods in Anthropology: Qualitative an Quantitative Approaches. Landham, MD: Altamira Press 2002.
- [Background] Atlas ti. Atlas.ti version 4.0 for Windows [computer program]. Version. Berlin, Germany. 1997.
- [Background] Friedemann-Sanchez G, Griffin JM, Partin MR. Gender differences in colorectal cancer screening barriers and information needs. Health Expect. 2007 Jun;10(2):148-60. doi: 10.1111/j.1369-7625.2006.00430.x. PMID 17524008
- [Background] Cooney NL, Litt MD, Cooney JL, Pilkey DT, Steinberg HR, Oncken CA. Concurrent brief versus intensive smoking intervention during alcohol dependence treatment. Psychol Addict Behav. 2007 Dec;21(4):570-5. doi: 10.1037/0893-164X.21.4.570. PMID 18072840
- [Background] Winer BJ. Statistical principles in experimental design (2nd Ed.). New York: McGraw-Hill; 1971.
- [Background] Little R, Rubin D. Statistical Analysis with Missing Data. 2nd ed. New York, NY: Wiley; 2002.
- [Background] Rubin D. Multiple Imputation for Non-Response in Surveys. New York: John Wiley & Sons, 1987.
- [Background] Brownson RC, Jones E. Bridging the gap: translating research into policy and practice. Prev Med. 2009 Oct;49(4):313-5. doi: 10.1016/j.ypmed.2009.06.008. Epub 2009 Jun 22. PMID 19555708
- [Background] Rogers EM. Diffusion of Innovations. New York: Free Press; 2003.
- [Result] Connor SE, Cook RL, Herbert MI, Neal SM, Williams JT. Smoking cessation in a homeless population: there is a will, but is there a way? J Gen Intern Med. 2002 May;17(5):369-72. doi: 10.1046/j.1525-1497.2002.10630.x. PMID 12047734
- [Result] Fischer PJ, Breakey WR. The epidemiology of alcohol, drug, and mental disorders among homeless persons. Am Psychol. 1991 Nov;46(11):1115-28. doi: 10.1037//0003-066x.46.11.1115. PMID 1772149
- [Result] Chau S, Chin M, Chang J, Luecha A, Cheng E, Schlesinger J, Rao V, Huang D, Maxwell AE, Usatine R, Bastani R, Gelberg L. Cancer risk behaviors and screening rates among homeless adults in Los Angeles County. Cancer Epidemiol Biomarkers Prev. 2002 May;11(5):431-8. PMID 12010856
- [Result] Torchalla I, Strehlau V, Okoli CT, Li K, Schuetz C, Krausz M. Smoking and predictors of nicotine dependence in a homeless population. Nicotine Tob Res. 2011 Oct;13(10):934-42. doi: 10.1093/ntr/ntr101. Epub 2011 May 26. PMID 21622493
- [Result] Mokdad AH, Marks JS, Stroup DF, Gerberding JL. Actual causes of death in the United States, 2000. JAMA. 2004 Mar 10;291(10):1238-45. doi: 10.1001/jama.291.10.1238. PMID 15010446
- [Result] Hwang SW, Lebow JM, Bierer MF, O'Connell JJ, Orav EJ, Brennan TA. Risk factors for death in homeless adults in Boston. Arch Intern Med. 1998 Jul 13;158(13):1454-60. doi: 10.1001/archinte.158.13.1454. PMID 9665356
- [Result] Barrow SM, Herman DB, Cordova P, Struening EL. Mortality among homeless shelter residents in New York City. Am J Public Health. 1999 Apr;89(4):529-34. doi: 10.2105/ajph.89.4.529. PMID 10191796
- [Result] Hwang SW. Mortality among men using homeless shelters in Toronto, Ontario. JAMA. 2000 Apr 26;283(16):2152-7. doi: 10.1001/jama.283.16.2152. PMID 10791509
- [Result] Kerker BD, Bainbridge J, Kennedy J, Bennani Y, Agerton T, Marder D, Forgione L, Faciano A, Thorpe LE. A population-based assessment of the health of homeless families in New York City, 2001-2003. Am J Public Health. 2011 Mar;101(3):546-53. doi: 10.2105/AJPH.2010.193102. Epub 2011 Jan 13. PMID 21233439
- [Result] Cousineau MR. Health status of and access to health services by residents of urban encampments in Los Angeles. J Health Care Poor Underserved. 1997 Feb;8(1):70-82. doi: 10.1353/hpu.2010.0378. PMID 9019027
- [Result] Hibbs JR, Benner L, Klugman L, Spencer R, Macchia I, Mellinger A, Fife DK. Mortality in a cohort of homeless adults in Philadelphia. N Engl J Med. 1994 Aug 4;331(5):304-9. doi: 10.1056/NEJM199408043310506. PMID 8022442
- [Result] HUD. Homelessness: Programs and the people they serve. Washington, DC: US Housing and Urban Development ; 1999
- [Result] Salit SA, Kuhn EM, Hartz AJ, Vu JM, Mosso AL. Hospitalization costs associated with homelessness in New York City. N Engl J Med. 1998 Jun 11;338(24):1734-40. doi: 10.1056/NEJM199806113382406. PMID 9624194
- [Result] Sachs-Ericsson N, Wise E, Debrody CP, Paniucki HB. Health problems and service utilization in the homeless. J Health Care Poor Underserved. 1999 Nov;10(4):443-52. doi: 10.1353/hpu.2010.0717. PMID 10581887
- [Result] Ferenchick GS. The medical problems of homeless clinic patients: a comparative study. J Gen Intern Med. 1992 May-Jun;7(3):294-7. doi: 10.1007/BF02598086. PMID 1613610
- [Result] Butler J, Okuyemi KS, Jean S, Nazir N, Ahluwalia JS, Resnicow K. Smoking characteristics of a homeless population. Subst Abus. 2002 Dec;23(4):223-31. doi: 10.1080/08897070209511495. PMID 12438835
- [Result] Wilder Foundation. Homeless Adults and Children in Minnesota Statewide Survey. 2004; http;//www.wilder.org/fileadmin/user upload/research/ Homeless2003/adult/StatewideAdultsByMetroGreaterMN Tables 192-199.pdf. Accessed September 29, 2006, 2006.
- [Result] Gelberg L, Linn LS. Demographic differences in health status of homeless adults. J Gen Intern Med. 1992 Nov-Dec;7(6):601-8. doi: 10.1007/BF02599198. PMID 1453243
- [Result] Kushel MB, Vittinghoff E, Haas JS. Factors associated with the health care utilization of homeless persons. JAMA. 2001 Jan 10;285(2):200-6. doi: 10.1001/jama.285.2.200. PMID 11176814
- [Result] Sees KL, Clark HW. When to begin smoking cessation in substance abusers. J Subst Abuse Treat. 1993 Mar-Apr;10(2):189-95. doi: 10.1016/0740-5472(93)90044-3. PMID 8510193
- [Result] Glassman AH. Cigarette smoking: implications for psychiatric illness. Am J Psychiatry. 1993 Apr;150(4):546-53. doi: 10.1176/ajp.150.4.546. PMID 8465868
- [Result] Hurt RD, Offord KP, Croghan IT, Gomez-Dahl L, Kottke TE, Morse RM, Melton LJ 3rd. Mortality following inpatient addictions treatment. Role of tobacco use in a community-based cohort. JAMA. 1996 Apr 10;275(14):1097-103. doi: 10.1001/jama.275.14.1097. PMID 8601929
- [Result] Burling TA, Ziff DC. Tobacco smoking: a comparison between alcohol and drug abuse inpatients. Addict Behav. 1988;13(2):185-90. doi: 10.1016/0306-4603(88)90010-x. PMID 3369328
- [Result] Hughes JR. Clinical implications of the association between smoking and alcoholism, in Alcohol and Tobacco: From basic science to policy: NIAAA Research Monograph 30. Washington, DC; US Government Printing Press; 1995
- [Result] Kozlowski LT, Skinner W, Kent C, Pope MA. Prospects for smoking treatment in individuals seeking treatment for alcohol and other drug problems. Addict Behav. 1989;14(3):273-8. doi: 10.1016/0306-4603(89)90058-0. PMID 2750568
- [Result] Anthony, JC., Warner, L A., & Kessler, RC.Comparative epidemiology of dependence on tobacco, alcohol, controlled substances, and inhalants: Basic findings from the National Comorbidity Survey. Experimental and Clinical Psychopharmacology, 2(3), 244-268. (1994).
- [Result] Chiolero A, Wietlisbach V, Ruffieux C, Paccaud F, Cornuz J. Clustering of risk behaviors with cigarette consumption: A population-based survey. Prev Med. 2006 May;42(5):348-53. doi: 10.1016/j.ypmed.2006.01.011. Epub 2006 Feb 28. PMID 16504277
- [Result] Falk DE, Yi HY, Hiller-Sturmhofel S. An epidemiologic analysis of co-occurring alcohol and tobacco use and disorders: findings from the National Epidemiologic Survey on Alcohol and Related Conditions. Alcohol Res Health. 2006;29(3):162-71. PMID 17373404
- [Result] Dawson DA. Drinking as a risk factor for sustained smoking. Drug Alcohol Depend. 2000 Jun 1;59(3):235-49. doi: 10.1016/s0376-8716(99)00130-1. PMID 10812284
- [Result] Kahler CW, Borland R, Hyland A, McKee SA, Thompson ME, Cummings KM. Alcohol consumption and quitting smoking in the International Tobacco Control (ITC) Four Country Survey. Drug Alcohol Depend. 2009 Mar 1;100(3):214-20. doi: 10.1016/j.drugalcdep.2008.10.006. Epub 2008 Dec 3. PMID 19056188
- [Result] McKee SA, Falba T, O'Malley SS, Sindelar J, O'Connor PG. Smoking status as a clinical indicator for alcohol misuse in US adults. Arch Intern Med. 2007 Apr 9;167(7):716-21. doi: 10.1001/archinte.167.7.716. PMID 17420431
- [Result] Castellsague X, Munoz N, De Stefani E, Victora CG, Castelletto R, Rolon PA, Quintana MJ. Independent and joint effects of tobacco smoking and alcohol drinking on the risk of esophageal cancer in men and women. Int J Cancer. 1999 Aug 27;82(5):657-64. doi: 10.1002/(sici)1097-0215(19990827)82:53.0.co;2-c. PMID 10417762
- [Result] Pelucchi C, Gallus S, Garavello W, Bosetti C, La Vecchia C. Cancer risk associated with alcohol and tobacco use: focus on upper aero-digestive tract and liver. Alcohol Res Health. 2006;29(3):193-8. PMID 17373408
- [Result] Schmidt W, Popham RE. The role of drinking and smoking in mortality from cancer and other causes in male alcoholics. Cancer. 1981 Mar 1;47(5):1031-41. doi: 10.1002/1097-0142(19810301)47:53.0.co;2-c. PMID 7226036
- [Result] Baca CT, Yahne CE. Smoking cessation during substance abuse treatment: what you need to know. J Subst Abuse Treat. 2009 Mar;36(2):205-19. doi: 10.1016/j.jsat.2008.06.003. Epub 2008 Aug 20. PMID 18715746
- [Result] Joseph A, Lexau B, Willenbring M, Nugent S, Nelson D. Factors associated with readiness to stop smoking among patients in treatment for alcohol use disorder. Am J Addict. 2004 Jul-Sep;13(4):405-17. doi: 10.1080/10550490490483116. PMID 15370939
- [Result] United States Department of health and Human Services, ed Treating Tobacco Use and Dependence. Washington, DC: U.S. Dept. of Health and Human Services, Public Health Service; 2008.
- [Result] Burling TA, Marshall GD, Seidner AL. Smoking cessation for substance abuse inpatients. J Subst Abuse. 1991;3(3):269-76. doi: 10.1016/s0899-3289(10)80011-2. PMID 1668228
- [Result] Hurt RD, Eberman KM, Croghan IT, Offord KP, Davis LJ Jr, Morse RM, Palmen MA, Bruce BK. Nicotine dependence treatment during inpatient treatment for other addictions: a prospective intervention trial. Alcohol Clin Exp Res. 1994 Aug;18(4):867-72. doi: 10.1111/j.1530-0277.1994.tb00052.x. PMID 7978097
- [Result] Bobo JK, McIlvain HE, Lando HA, Walker RD, Leed-Kelly A. Effect of smoking cessation counseling on recovery from alcoholism: findings from a randomized community intervention trial. Addiction. 1998 Jun;93(6):877-87. doi: 10.1046/j.1360-0443.1998.9368779.x. PMID 9744123
- [Result] Gariti P, Alterman A, Mulvaney F, Mechanic K, Dhopesh V, Yu E, Chychula N, Sacks D. Nicotine intervention during detoxification and treatment for other substance use. Am J Drug Alcohol Abuse. 2002 Nov;28(4):671-9. doi: 10.1081/ada-120015875. PMID 12492263
- [Result] Kalman D, Hayes K, Colby SM, Eaton CA, Rohsenow DJ, Monti PM. Concurrent versus delayed smoking cessation treatment for persons in early alcohol recovery. A pilot study. J Subst Abuse Treat. 2001 Apr;20(3):233-8. doi: 10.1016/s0740-5472(00)00174-4. PMID 11516593
- [Result] Cooney NL, Litt MD, Cooney JL, Pilkey DT, Steinberg HR, Oncken CA. Alcohol and tobacco cessation in alcohol-dependent smokers: analysis of real-time reports. Psychol Addict Behav. 2007 Sep;21(3):277-86. doi: 10.1037/0893-164X.21.3.277. PMID 17874878
- [Result] Schneider NG. Nicotine therapy in smoking cessation. Pharmacokinetic considerations. Clin Pharmacokinet. 1992 Sep;23(3):169-72. doi: 10.2165/00003088-199223030-00001. No abstract available. PMID 1511534
- [Result] Cooney NL, Cooney JL, Perry BL, Carbone M, Cohen EH, Steinberg HR, Pilkey DT, Sevarino K, Oncken CA, Litt MD. Smoking cessation during alcohol treatment: a randomized trial of combination nicotine patch plus nicotine gum. Addiction. 2009 Sep;104(9):1588-96. doi: 10.1111/j.1360-0443.2009.02624.x. Epub 2009 Jun 22. PMID 19549054
- [Result] Cooney JL, Cooney NL, Patten Ca, George TP. Comorbidity of Nicotine Dependence with affective, psychotic and substance treatment disorders. New York: Marcel Dekker; 2004.
- [Result] Istvan J, Matarazzo JD. Tobacco, alcohol, and caffeine use: a review of their interrelationships. Psychol Bull. 1984 Mar;95(2):301-26. No abstract available. PMID 6544436
- [Result] Monti PM, Rohsenow DJ, Colby Sm, Abrams DB. Smoking among alcoholics during and after treatment: implications for models, treatment strategies, and policy.In Fertig JB, Allen JP, eds. alcohol and tobacco: from basic science to clinical practice. Vol NIH pub. No. 95-3931. Bethesda, MD: National Institute of Health, National institute on Alcohol Abuse and Alcoholism; 1995
- [Result] Cooney JL, Cooney NL, Pilkey DT, Kranzler HR, Oncken CA. Effects of nicotine deprivation on urges to drink and smoke in alcoholic smokers. Addiction. 2003 Jul;98(7):913-21. doi: 10.1046/j.1360-0443.2003.00337.x. PMID 12814497
- [Result] Palfai TP, Monti PM, Ostafin B, Hutchison K. Effects of nicotine deprivation on alcohol-related information processing and drinking behavior. J Abnorm Psychol. 2000 Feb;109(1):96-105. doi: 10.1037//0021-843x.109.1.96. PMID 10740940
- [Result] Muraven M, Baumeister RF. Self-regulation and depletion of limited resources: does self-control resemble a muscle? Psychol Bull. 2000 Mar;126(2):247-59. doi: 10.1037/0033-2909.126.2.247. PMID 10748642
- [Result] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Result] Babor TF, Higgins-Biddle JC, Saunders JB, Monteiro MG. AUDIT: The alcohol Use Disorders Identification Test-Guidelines for Use in Primary Care. Second Edition. Geneva Switzerland: world Health Organization, Department of Mental Health and Substance Abuse Dependence; 2001.
- [Result] Bech P, Larsen JK, Andersen J. The BPRS: psychometric developments. Psychopharmacol Bull. 1988;24(1):118-21. No abstract available. PMID 3387515
- [Result] Raskin A. Discussion: recent developments in ascertainment and scaling of the BPRS. Psychopharmacol Bull. 1988;24(1):122-4. No abstract available. PMID 3387516
- [Result] Roncone R, Ventura J, Impallomeni M, Falloon IR, Morosini PL, Chiaravalle E, Casacchia M. Reliability of an Italian standardized and expanded Brief Psychiatric Rating Scale (BPRS 4.0) in raters with high vs. low clinical experience. Acta Psychiatr Scand. 1999 Sep;100(3):229-36. doi: 10.1111/j.1600-0447.1999.tb10850.x. PMID 10493090
- [Result] Ruggeri M, Koeter M, Schene A, Bonetto C, Vazquez-Barquero JL, Becker T, Knapp M, Knudsen HC, Tansella M, Thornicroft G; EPSILON Study Group. Factor solution of the BPRS-expanded version in schizophrenic outpatients living in five European countries. Schizophr Res. 2005 Jun 1;75(1):107-17. doi: 10.1016/j.schres.2004.05.017. PMID 15820329
- [Result] Goldade K, Choi K, Bernat DH, Klein EG, Okuyemi KS, Forster J. Multilevel predictors of smoking initiation among adolescents: findings from the Minnesota Adolescent Community Cohort (MACC) study. Prev Med. 2012 Mar-Apr;54(3-4):242-6. doi: 10.1016/j.ypmed.2011.12.029. Epub 2012 Jan 8. PMID 22245269
- [Result] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Result] Hajek P, West R, Foulds J, Nilsson F, Burrows S, Meadow A. Randomized comparative trial of nicotine polacrilex, a transdermal patch, nasal spray, and an inhaler. Arch Intern Med. 1999 Sep 27;159(17):2033-8. doi: 10.1001/archinte.159.17.2033. PMID 10510989
- [Result] Orleans CT, Resch N, Noll E, Keintz MK, Rimer BK, Brown TV, Snedden TM. Use of transdermal nicotine in a state-level prescription plan for the elderly. A first look at 'real-world' patch users. JAMA. 1994 Feb 23;271(8):601-7. PMID 8301792
- [Result] Jolicoeur DG, Ahluwalia JS, Richter KP, Mosier M, Harris KJ, Gibson C, Moranetz CA. The use of nicotine patches with minimal intervention. Prev Med. 2000 Jun;30(6):504-12. doi: 10.1006/pmed.2000.0670. PMID 10901493
- [Result] Allen JO, Wilson VB, eds. Assessing Alcohol Problems: a Guide for Clinicians and Researchers. Second Ed. Bethesda. Maryland, USA: U.S. Department of Health and Human Services. Public Health Service. National Institute on Alcohol Abuse and Alcoholism; 2003; No. NIH Publication NO. 03-3745.
- [Result] Shelley D, Cantrell J, Wong S, Warn D. Smoking cessation among sheltered homeless: a pilot. Am J Health Behav. 2010 Sep-Oct;34(5):544-52. doi: 10.5993/ajhb.34.5.4. PMID 20524884
- [Result] Kadden R, Carroll K, Donovan D, Cooney N, Monti P, Abrams D. et al. Cognitive-Behavioral coping skills therapy Manual: Clinical research Guide for therapist cognitive- behavioral coping skills Therapy Manual: a clinical research guide for therapists counseling patients with alcohol abuse and dependence. Vol 3. DHHS publication no. (ADM) 92-1895 ed. Rockville, MD: US Government Printing Office; 1992.
- [Result] Babor TF, Higgins-Biddle JC. Alcohol screening and brief intervention: dissemination strategies for medical practice and public health. Addiction. 2000 May;95(5):677-86. doi: 10.1046/j.1360-0443.2000.9556773.x. PMID 10885042
- [Result] Guiterrez-Bedmar M, Segui-Gomez M, Gomez-Gracia E, Bes-Rastrollo M, Martinez-Gonzalez MA. Smoking status, changes in smoking status and health-related quality of life: findings from the SUN ("Seguimiento Universidad de Navarra") cohort. Int J Environ Res Public Health. 2009 Jan;6(1):310-20. doi: 10.3390/ijerph6010310. Epub 2009 Jan 19. PMID 19440285
- [Result] Sarna L, Bialous SA, Cooley ME, Jun HJ, Feskanich D. Impact of smoking and smoking cessation on health-related quality of life in women in the Nurses' Health Study. Qual Life Res. 2008 Dec;17(10):1217-27. doi: 10.1007/s11136-008-9404-8. Epub 2008 Oct 18. PMID 18931942
- [Result] Williams MV, Parker RM, Baker DW, Parikh NS, Pitkin K, Coates WC, Nurss JR. Inadequate functional health literacy among patients at two public hospitals. JAMA. 1995 Dec 6;274(21):1677-82. PMID 7474271
- [Result] SRNT Subcommittee on Biochemical Verification. Biochemical verification of tobacco use and cessation. Nicotine Tob Res. 2002 May;4(2):149-59. doi: 10.1080/14622200210123581. No abstract available. PMID 12028847
- [Result] Sobell L, Sobell M. Timeline follow-back: a technique for assessing self-reporting alcohol consumption In:. Timeline following-back: a technique for assessing self-reported alcohol consumption in:. Totowa, NJ: Humana Press; 1992.
- [Result] Miller WR, Del Boca FK. Measurement of drinking behavior using the Form 90 family of instruments. J Stud Alcohol Suppl. 1994 Dec;12:112-8. doi: 10.15288/jsas.1994.s12.112. PMID 7722987
- [Result] Goldade K, Whembolua GL, Thomas J, Eischen S, Guo H, Connett J, Des Jarlais D, Resnicow K, Gelberg L, Owen G, Grant J, Ahluwalia JS, Okuyemi KS. Designing a smoking cessation intervention for the unique needs of homeless persons: a community-based randomized clinical trial. Clin Trials. 2011 Dec;8(6):744-54. doi: 10.1177/1740774511423947. PMID 22167112
- [Result] Okuyemi KS, Thomas JL, Hall S, Nollen NL, Richter KP, Jeffries SK, Caldwell AR, Ahluwalia JS. Smoking cessation in homeless populations: a pilot clinical trial. Nicotine Tob Res. 2006 Oct;8(5):689-99. doi: 10.1080/14622200600789841. PMID 17008196
- [Result] Fagerstrom KO. Measuring degree of physical dependence to tobacco smoking with reference to individualization of treatment. Addict Behav. 1978;3(3-4):235-41. doi: 10.1016/0306-4603(78)90024-2. No abstract available. PMID 735910
- [Result] Hughes JR, Hatsukami D. Signs and symptoms of tobacco withdrawal. Arch Gen Psychiatry. 1986 Mar;43(3):289-94. doi: 10.1001/archpsyc.1986.01800030107013. PMID 3954551
- [Result] Shiffman S, West R, Gilbert D; SRNT Work Group on the Assessment of Craving and Withdrawal in Clinical Trials. Recommendation for the assessment of tobacco craving and withdrawal in smoking cessation trials. Nicotine Tob Res. 2004 Aug;6(4):599-614. doi: 10.1080/14622200410001734067. PMID 15370156
- [Result] Cox LS, Tiffany ST, Christen AG. Evaluation of the brief questionnaire of smoking urges (QSU-brief) in laboratory and clinical settings. Nicotine Tob Res. 2001 Feb;3(1):7-16. doi: 10.1080/14622200020032051. PMID 11260806
- [Result] Flannery BA, Roberts AJ, Cooney N, Swift RM, Anton RF, Rohsenow DJ. The role of craving in alcohol use, dependence, and treatment. Alcohol Clin Exp Res. 2001 Feb;25(2):299-308. PMID 11236847
- [Derived] Pratt R, Xiong S, Kmiecik A, Strobel-Ayres C, Joseph A, Rose SAE, Luo X, Cooney N, Thomas J, Specker S, Okuyemi K. The implementation of a smoking cessation and alcohol abstinence intervention for people experiencing homelessness. BMC Public Health. 2022 Jun 27;22(1):1260. doi: 10.1186/s12889-022-13563-5. PMID 35761310
- [Derived] Pratt R, Pernat C, Kerandi L, Kmiecik A, Strobel-Ayres C, Joseph A, Everson Rose SA, Luo X, Cooney N, Thomas J, Okuyemi K. "It's a hard thing to manage when you're homeless": the impact of the social environment on smoking cessation for smokers experiencing homelessness. BMC Public Health. 2019 May 24;19(1):635. doi: 10.1186/s12889-019-6987-7. PMID 31126265
- [Derived] Ojo-Fati O, Joseph AM, Ig-Izevbekhai J, Thomas JL, Everson-Rose SA, Pratt R, Raymond N, Cooney NL, Luo X, Okuyemi KS. Practical issues regarding implementing a randomized clinical trial in a homeless population: strategies and lessons learned. Trials. 2017 Jul 5;18(1):305. doi: 10.1186/s13063-017-2046-9. PMID 28679430
- [Derived] Ojo-Fati O, John F, Thomas J, Joseph AM, Raymond NC, Cooney NL, Pratt R, Rogers CR, Everson-Rose SA, Luo X, Okuyemi KS. Integrating smoking cessation and alcohol use treatment in homeless populations: study protocol for a randomized controlled trial. Trials. 2015 Aug 29;16:385. doi: 10.1186/s13063-015-0858-z. PMID 26320081

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Integrated Intensive Smoking + Alcohol | Usual Care
Started | 172 | 180
Completed | 170 | 180
Not Completed | 2 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Intensive Smoking + Alcohol | Usual Care | Total
Number analyzed (Participants) | 172 | 180 | 352
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 167 | 175 | 342
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (10.6) | 46 (11.3) | 46 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 48 | 76
  Male | 144 | 132 | 276
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 5 | 6
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 127 | 123 | 250
  White | 28 | 32 | 60
  More than one race | 8 | 14 | 22
  Unknown or Not Reported | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: CO-verified Smoking Status at 26 Weeks
Description: Smoking status is verified by measuring the concentration of carbon monoxide (CO) in expired air. Participants with a breath CO content less than or equal to 8 parts per million are characterized as abstinent from smoking for at least 7 days.
Time Frame: 7-day smoking abstinence at week 26 follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Integrated Intensive Smoking + Alcohol | Usual Care
Number analyzed (Participants) | 172 | 180
percentage of participants | 16.3 | 12.6

2. Secondary Outcome: CO-verified Smoking Status at 12 Weeks
Description: as for outcome 1
Time Frame: at weeks 12
Measure: Number; unit: percentage of participants
Arm/Group | Integrated Intensive Smoking + Alcohol | Usual Care
Number analyzed (Participants) | 172 | 180
percentage of participants | 21.6 | 14

3. Other Pre Specified Outcome: Self-Reported Continuous Alcohol Abstinence for 30 Days
Description: Participants will use a self-administered timeline-followback instrument, which asks them to retrospectively estimate their alcohol use in the 30 days prior to the report date. Outcome is reported as the mean number of continuous alcohol-free days over the past 30 day period.
Time Frame: at week 26
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Integrated Intensive Smoking + Alcohol | Usual Care
Number analyzed (Participants) | 172 | 180
days | 3.4 (.71) | 3.9 (.71)

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Integrated Intensive Smoking + Alcohol | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/172 | 1/180
Serious Adverse Events (participants affected / at risk) | 0/172 | 0/180
Other Adverse Events (participants affected / at risk) | 90/172 | 101/180
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Integrated Intensive Smoking + Alcohol (N=172) | Usual Care (N=180)
Addiction Services (Psychiatric disorders) | 0 (0) | 2 (2)
Allergy (Immune system disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2)
Breathing Difficulties (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1)
Dental Pain (General disorders) | 2 (2) | 4 (4)
Depression (Psychiatric disorders) | 3 (4) | 1 (1)
Diabetes (Endocrine disorders) | 4 (4) | 0 (0)
Eye Irritation (Eye disorders) | 1 (1) | 0 (0)
Fainting (General disorders) | 3 (3) | 1 (1)
Flu-Like Symptoms (General disorders) | 3 (3) | 0 (0)
Foot Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Frostbite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Gastrointestinal Issues (Gastrointestinal disorders) | 6 (6) | 4 (4)
Gynecological Issues (Reproductive system and breast disorders) | 2 (2) | 2 (3)
Headache (General disorders) | 2 (2) | 2 (3)
Heart Problems (Cardiac disorders) | 2 (2) | 1 (1)
High Blood Pressure (Cardiac disorders) | 2 (2) | 4 (4)
Infection (Infections and infestations) | 5 (5) | 9 (10)
Injury (Injury, poisoning and procedural complications) | 9 (10) | 15 (17)
Medication Review (General disorders) | 4 (4) | 2 (2)
NRT Patch Irritation (Skin and subcutaneous tissue disorders) | 7 (8) | 21 (22) — Nicotine Replacement Therapy (NRT)
Pain (General disorders) | 10 (11) | 10 (12)
Seizure (Nervous system disorders) | 0 (0) | 3 (5)
Suicidality (Psychiatric disorders) | 2 (4) | 0 (0)
Surgery (Surgical and medical procedures) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT01932996/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT01932996/ICF_001.pdf